CLINICAL TRIAL: NCT01074606
Title: Visual Function After Implantation of AcrySof® Toric Lens
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated based on a business decision.
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-0902
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2011-08

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toric (Experimental): AcrySof Toric Intraocular Lens (IOL)
  Interventions: Device: AcrySof Toric Intraocular Lens

INTERVENTIONS:
Device: AcrySof Toric Intraocular Lens — Implantation of the AcrySof Toric Intraocular Lens (IOL)

SUMMARY:
The objective of this study is to evaluate the postoperative visual function of Taiwanese patients following bilateral or unilateral AcrySof Toric Intraocular Lens (IOL) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Prospective subjects should be adults and may be of any race and gender, and diagnosed with cataracts.
* Subject must require extraction of cataracts followed by implantation of a posterior chamber intraocular lens.
* All subjects must have between 0.75 - 2.0 Diopter (D) of astigmatism preoperatively as measured by keratometry readings.
* For any second eye surgery in bilateral AcrySof Toric patients, it should be performed at least one week following the first eye implant but no longer than one month after the first implant.

Exclusion Criteria:

* Subjects with pre-existing conditions that could skew the results should be excluded from the Study.
* AcrySof® Toric product inserts under "Precautions" for subject groups that should be excluded from this Study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Refractive Cylinder | Pre-Operative Day, 1 Month Postoperative, 3 Month Postoperative

SECONDARY OUTCOMES:
Uncorrected distance visual acuity (UCDVA) | Pre-Operative Day, 1 Month Postoperative, 3 Month Postoperative
Best corrected distance visual acuity (BDCVA) | Pre-operative, 1 month postoperative, 3 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua, Taiwan